CLINICAL TRIAL: NCT06599710
Title: Pilot Study to Evaluate the Effects of a Food Product Containing Mushroom Extracts (AndosanTM) in Subjects with Colorectal Cancer-Related Fatigue
Brief Title: The Effects of a Food Product Containing Mushroom Extracts (AndoSanTM) in Subjects with Colorectal Cancer-related Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mycotech Pharma AS (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BTS2088/24
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cancer-related Fatigue
Keywords: Cancer-related fatigue; Colorectal cancer; Andosan; Agaricus blazei Murill; Hericium erinaceus; Agaricus subrufesence; Mushroom extract; Grifola frondosa; Chronic inflammation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm pilot nutritional study, multicentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AndoSan 6 week intervention (Other): Intervention; AndoSanTM, 60 ml/day for 6 weeks
  Interventions: Dietary Supplement: AndoSanTM

INTERVENTIONS:
Dietary Supplement: AndoSanTM — Fermented water-based exctract of Agaricus subrufesence, Hericum erinacus, and Grifola frondosa

SUMMARY:
Effects of a food product containing mushroom extracts (AndoSanTM) in subjects with colorectal cancer-related fatigue.

AndoSanTM is a specialized liquid food product that includes fermented extracts from the fungi Agaricus subrufesence (Agaricus blazei Murill), Hericium erinaceus, and Grifola frondosa as the main ingredients.

The primary study objective is to assess the change in complaints about cancer-related fatigue while taking AndoSanTM. Further objectives are to evaluate the change in health-related quality of life (QoL) and levels

DETAILED DESCRIPTION:
Pilot study to evaluate the effects of a food product containing mushroom extracts (AndoSanTM) in subjects with colorectal cancer-related fatigue.

AndoSanTM is a specialized liquid food product that includes fermented extracts from the fungi Agaricus subrufesence (Agaricus blazei Murill), Hericium erinaceus, and Grifola frondosa as the main ingredients.

The primary study objective is to assess the change in complaints related to cancer-related fatigue while taking AndoSanTM. Further objectives are to evaluate the change in health-related quality of life (QoL) and levels of inflammation markers, as well as its safety and tolerability while taking AndoSanTM.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females from 18 to 65 years of age
2. Caucasian
3. Diagnosis of non-metastatic colorectal cancer (stages I-III) (documented)
4. Diagnosis of persistent cancer-related fatigue with moderate or severe symptoms of cancer-related fatigue (≥ 4 on 0-10 Numerical Rating Scale (NRS) and a Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Fatigue subscale (FACIT-F FS) score of ≤ 34 for assessment of average fatigue in the week before visit 1, both assessed at visit 1)
5. Cancer-related fatigue present since at least 4 weeks before visit one at a stable level (self-reported)
6. Cancer treatment completed (as reported by the attending physician before the study) considering the following conditions:

   * a minimum of 4 weeks after the end of the last cancer-related therapy (e.g. chemotherapy, radiotherapy)
   * a minimum of 6 weeks after any cancer-related surgery (if any)
7. Serum C-reactive protein (CRP) levels greater than 3 mg/l at visit1/ Screening
8. Stable medication for comorbidities (if any)
9. Established cancer-related fatigue management regime in line with current guidelines, if any, since at least 4 weeks (e.g., physical exercise counseling, medication/supplementation, nutritional counseling, psychosocial counseling)
10. Expectedly to keep level of activity (including e.g. work/educational activities, physical activity) and dietary habits during the study, including caffeine consumption and liquid intake
11. Negative pregnancy test at V1 and willingness to use a reliable method of contraception during the study in women of childbearing potential
12. Readiness and ability to understand and comply with study requirements as judged by the investigator (to take the IP as recommended)

Exclusion Criteria

1. Rapidly progressing cancer without reasonable treatment options and/or serious worsening of cancer disease during the study, as well as the need for any cancer treatment that expectedly may need to start and/or cancer-related fatigue management that expectedly may need to start/get modified during the study
2. Severe anemia (hemoglobin (Hb) ≤ 8 g/dl within last 2 weeks before or at visit 1
3. Acute illness or uncontrolled chronic metabolic illness (including diabetes mellitus, hyperthyroidism, hypothyroidism, and excluding adequately medicated hypothyroidism), uncontrolled pain, and other disorders known to cause fatigue complaints (such as heart failure, chronic obstructive pulmonary disease (COPD), severe deconditioning and/or sarcopenia, severe and unresponsive inflammation, severe damage of gastrointestinal organs impairing oral food intake and digestion, parenteral nutrition, decreased calorie intake due to substantial appetite loss), all as per investigator's judgment
4. Psychiatric disorders, including recently occurred (within the last 12 weeks before visit 1) or severe depression as judged by the investigator (stable treatment with low-dose selective serotonin reuptake inhibitors (SSRIs) is permitted)
5. Known HIV infection, hepatitis B or C, or active tuberculosis (self-reported)
6. Major surgery within 4 weeks before study or planned surgery during the treatment period
7. Consuming any other food supplements / FSMPs during the study, e.g. ginseng, guarana, mistletoe
8. History of or current abuse of medication, e.g. opioids, drugs, or alcohol
9. Participation in another study during the last 30 days before and during the study
10. Breastfeeding
11. Any other reason for exclusion as per the investigator's judgment, e.g. hypersensitivity or allergy to the IP, (expected) insufficient compliance with study procedures (due to substantial cognitive complaints related to cancer-related fatigue or other cause)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Difference in the level of cancer-related fatigue after 6 weeks IP intake, in comparison to the baseline. | 6 weeks
  Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Fatigue Subscale (FS): The FACIT-F FS is a subscale that measures the level of fatigue in patients, particularly those with chronic illnesses like cancer. The subscale consists of a set of questions scored on a scale from 0 to 52, with higher scores indicating less fatigue and therefore a better outcome. A score of 0 would indicate severe fatigue, while a score of 52 reflects minimal to no fatigue.

SECONDARY OUTCOMES:
Further difference in the level of cancer-related fatigue after 6 weeks IP intake, in comparison to the baseline. | 6 weeks
  The difference in cancer-related fatigue after 3 weeks and after 6 weeks, each in comparison to the baseline: Cancer-related fatigue is assessed using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Fatigue Subscale (FS). This scale ranges from 0 to 52, where higher scores indicate a better outcome.
  The differences in health-related Quality of Life (QoL) using the FACIT-F subscales relating to physical, social/family, emotional, and functional well-Health-related QoL is measured using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) subscales, which cover physical, social/family, emotional, and functional well-being. Each subscale has its own scoring range (typically 0 to 28) where higher scores indicate a better outcome.
  The analysis compares fatigue levels at 3 and 6 weeks to the baseline, with changes in scores reflecting either improvement or worsening of fatigue symptoms over time.

OTHER OUTCOMES:
The difference in the levels of inflammation markers (serum/plasma) after 3 weeks and after 6 weeks, each in comparison to the baseline. | 6 weeks
  Measurement of inflammation related parameters in blood; CRP, IL-1ß, IL-1 RA, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-17A, INF-gamma, TNF-alpha.
  The difference in gut microbiome profiles and calprotectin levels before and after 6 weeks of IP intake.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - BioTeSys GmbH, Esslingen am Neckar, Baden-Wurttemberg
  - BioTeSys, Esslingen am Neckar, Baden-Wurttemberg
  - analyze & realize GmbH, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No
Data might not be shared due to intellectual property concerns.